CLINICAL TRIAL: NCT01343381
Title: Anticoagulant Effect and Reversal of Hepalean Compared With PPC Heparin in Patients Undergoing Cardiopulmonary Bypass: a Pilot Randomized Trial
Brief Title: Comparison of Heparin Types; Efficacy and Safety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CANNeCTIN
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Disease
Keywords: Heparin; Coronary artery bypass graft surgery; Anti-coagulation efficacy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepalean Heparin (Active Comparator)
  Interventions: Drug: Hepalean Heparin
- PPC Heparin (Active Comparator)
  Interventions: Drug: PPC Heparin

INTERVENTIONS:
Drug: Hepalean Heparin — 400 units per kilogram bolus prior to initiation of CPB
  Arms: Hepalean Heparin
Drug: PPC Heparin — 400 unit per kilogram bolus prior to initiation of CPB
  Arms: PPC Heparin

SUMMARY:
Heparin, a blood thinner, is used routinely in Open-heart surgery. Do different brands of this drug have differing clinical effects despite both having exactly the same regulation and marketing specifications?

ELIGIBILITY:
Inclusion Criteria:

* will be undergoing cardiopulmonary bypass for coronary artery disease
* has provided written informed consent

Exclusion Criteria:

* Allergy or intolerance to Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Feasibility to conduct a larger trial | pre-cardiopulmonary bypass initiation; peri-operative period (in minutes) to 24 hours post-operatively
  Will the pilot show that the pilot's design is feasible with respect to timely patient enrolment, blinding of treatment allocation, study drug dosage requirements and the collection and measurement of study outcomes; ACT of > 450 seconds after initial pre-CPB heparin bolus, dosage of additional heparin (if any) to maintain an ACT of greater than 450 seconds, differences (if any) in coagulation profiles, differences if any in chest tube drainage, differences (if any) in post-operative transfusion requiements

SECONDARY OUTCOMES:
ACT after initial dose of heparin | pre-cardiopulmonary bypass initiation; peri-operatively(in seconds)
  A dose of 400 units/kgm will be used
Total Heparin Dose used | pre-cardiopulmonary bypass initiation to termination of cardiopulmonary bypass; peri-operatively(in minutes)
  The total dose of heparin needed to maintain an ACT of 480 seconds throught bypass time.
Coagulation | post-cardiopulmonary inition, at the 45 minute on pump time point; perioperatively to 24 hours post-operatively
  aPTT, TCT, anti-Xa and anti IL IIa activity ant TAT levels after initial heparin dose and after 45 minutes on CPB.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin H Teoh, MD, Principal Investigator — Hamilton Health Sciences: Hamilton General Site
Locations (1):
- Hamilton Health Sciences: Hamilton General Hospital, Hamilton, Ontario, Canada